CLINICAL TRIAL: NCT01226485
Title: A Phase 1 Dose-Escalation Study of LY2940680 in Patients With Advanced Cancer
Brief Title: A Study in Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lilly 13200; I4J-MC-HHBB (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Advanced Cancer
Keywords: Cancer; Terminal; Solid Tumor; End Stage; Metastatic
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — LY2940680

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Taladegib (Experimental): Part A Cohort 1: 50 milligram (mg) taladegib administered orally QD on a 28-day cycle.
  Part A Cohort 2: 100 mg taladegib administered orally QD on a 28-day cycle.
  Part A Cohort 3: 200 mg taladegib administered orally QD on a 28-day cycle.
  Part A Cohort 4: 400 mg taladegib administered orally QD on a 28-day cycle.
  Part A Cohort 5: 600 mg taladegib administered orally QD on a 28-day cycle.
  Part C: 400 mg taladegib administered orally QD. Participants with advanced solid tumors.
  Part D: 400 mg taladegib administered orally QD. Participants with advanced basal cell carcinoma (BCC).
  Interventions: Drug: Taladegib

INTERVENTIONS:
Drug: Taladegib — Administered IV
  Other Names: LY2940680

SUMMARY:
The purpose of this study is to find a recommended dose level and schedule of dosing LY2940680 that can safely be taken by participants with advanced cancer. The study will also explore the changes in a cancer marker level in skin, hair follicles, buccal cells, and tumor cells. Finally, the study will help document any antitumor activity this drug may have.

DETAILED DESCRIPTION:
Participants may include those who have previously received treatment with another hedgehog smoothened (Hh/Smo) inhibitor (excluding LY2940680).

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological evidence of a diagnosis of cancer that is advanced and/or metastatic. The patient must be, in the judgment of the investigator, an appropriate candidate for experimental therapy.
* Have the presence of measurable or nonmeasurable disease
* Have adequate organ function, including:

  * Hematologic: Absolute neutrophil count (ANC) greater than or equal to 1.5 x 109/L, platelets greater than or equal to 100 x 109/L, and hemoglobin greater than or equal to 9 g/dL. Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin until 5 days after the erythrocyte transfusion.
  * Hepatic: Bilirubin less than or equal to 1.5 times upper limits of normal (ULN), ALT, and aspartate transferase (AST) less than or equal to 2.0 times ULN. If the liver has tumor involvement AST and ALT equaling less than or equal to 5 times ULN are acceptable.
  * Renal: Serum creatinine less than or equal to 1.5 times ULN.
* Have a performance status of less than or equal to 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued previous treatments for cancer and recovered from the acute effects of therapy (for example, at least 42 days for mitomycin-C or nitrosoureas, 28 days for other chemotherapy and biologics. At the discretion of the investigator, hormone refractory prostate cancer patients who are stable on gonadotropin-releasing hormone (GnRH) agonist therapy and breast cancer patients who are stable on antiestrogen therapy (for example, an aromatase inhibitor) may continue treatment

Exclusion Criteria:

* Have received treatment within 21 days of the initial dose of study drug with an experimental agent for noncancer indications that has not received regulatory approval for any indication.
* Have serious preexisting medical conditions
* Have symptomatic central nervous system (CNS) malignancy (with the exception of medulloblastoma) or metastasis (screening not required). Patients with treated CNS metastases are eligible for this study if they are not currently receiving corticosteroids and/or anticonvulsants, and their disease is asymptomatic and radiographically stable for at least 60 days.
* Have known current hematologic malignancies or acute or chronic leukemia
* Have a known active fungal, bacterial, and/or known viral infection including human immunodeficiency (HIV) or viral (A, B, or C) hepatitis (screening is not required)
* Have a second primary malignancy that in the judgment of the investigator and sponsor may affect the interpretation of results
* Have QTc interval of >500 msec on screening electrocardiogram
* Patients who have previously received treatment with LY2940680

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-09; Primary Completion 2015-01 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- United States (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Redwood City, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Worth, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study completers are participants who received at least one dose of study drug and were evaluated for safety. Part B of the study was not implemented as the estimated half-life was considered long enough for once a day (QD) dosing.
Groups:
- Part A: Cohort 1: Part A Cohort 1: 50 milligram (mg) taladegib administered orally QD on a 28-day cycle.
- Part A: Cohort 2: Part A Cohort 2: 100 mg taladegib administered orally QD on a 28-day cycle.
- Part A: Cohort 3: Part A Cohort 3: 200 mg taladegib administered orally QD on a 28-day cycle.
- Part A: Cohort 4: Part A Cohort 4: 400 mg taladegib administered orally QD on a 28-day cycle.
- Part A: Cohort 5: Part A Cohort 5: 600 mg taladegib administered orally QD on a 28-day cycle.
- Part C: Part C: 400 mg taladegib administered orally QD. Participants with advanced solid tumors.
- Part D: Part D: 400 mg taladegib administered orally QD. Participants with advanced basal cell carcinoma (BCC).
Period: Overall Study
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Part A: Cohort 3 | Part A: Cohort 4 | Part A: Cohort 5 | Part C | Part D
Started | 3 | 6 | 3 | 6 | 7 | 19 | 40
Received at Least One Dose of Drug | 3 | 6 | 3 | 6 | 7 | 19 | 40
Completed | 3 | 6 | 3 | 6 | 7 | 19 | 40
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Part A: Cohort 2: Part A Cohort 2 : 100 mg taladegib administered orally QD on a 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Part A: Cohort 3 | Part A: Cohort 4 | Part A: Cohort 5 | Part C | Part D | Total
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 7 | 19 | 40 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (14.57) | 57.2 (14.18) | 67.3 (7.37) | 60.7 (14.05) | 65.6 (11.34) | 62.5 (10.59) | 64.0 (12.47) | 63.1 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 3 | 2 | 6 | 8 | 23
  Male | 2 | 4 | 2 | 3 | 5 | 13 | 32 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 4
  Not Hispanic or Latino | 3 | 6 | 2 | 6 | 7 | 18 | 38 | 80
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  White | 3 | 6 | 3 | 6 | 7 | 18 | 36 | 79
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 6 | 3 | 6 | 7 | 19 | 40 | 84

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose: Maximum Tolerated Dose
Description: Recommended Phase 2 dose was determined by maximum tolerated dose (MTD), which was determined by Dose-limiting toxicity (DLT). For the purpose of this study, the MTD was defined as the highest tested dose that had <33% probability of causing a DLT in Cycle 1 of Part A.
Time Frame: Time to First Dose to the End of Cycle 1 of Part A (Up To 28 Days)
Population: Part A participants who received at least one dose of study drug.
Measure: Number; unit: milligrams (mg)
Groups:
- All Part A Participants: Part A: Cohort 1 Part A Cohort 1: 50 milligram (mg) taladegib administered orally QD on a 28-day cycle.
  Part A: Cohort 2 Part A Cohort 2: 100 mg taladegib administered orally QD on a 28-day cycle.
  Part A: Cohort 3 Part A Cohort 3: 200 mg taladegib administered orally QD on a 28-day cycle.
  Part A: Cohort 4 Part A Cohort 4: 400 mg taladegib administered orally QD on a 28-day cycle.
  Part A: Cohort 5 Part A Cohort 5: 600 mg taladegib administered orally QD on a 28-day cycle.
Arm/Group | All Part A Participants
Number analyzed (Participants) | 25
milligrams (mg) | 400

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞])
Description: Pharmacokinetics (PK): 1.Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞])
Time Frame: Cycle 1, Day 1: Predose, 0.5, 1, 2, 4, 6, 8, 10,11, 12 hour(h), Day 15: Predose, 0.5, 1, 2, 4, 6, 8, 10,11, 12 h
Population: All participants who received at least one dose of study drug and had evaluable PK data. All participants who received 400 mg taladegib were analyzed together.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (μg*h/mL)
Groups:
- 50 mg Taladegib: 50 milligram (mg) taladegib administered orally QD on a 28-day cycle.
- 100 mg Taladegib: 100 mg taladegib administered orally QD on a 28-day cycle.
- 200 mg Taladegib: 200 mg taladegib administered orally QD on a 28-day cycle.
- 400 mg Taladegib: 400 mg taladegib administered orally QD on a 28-day cycle.
- 600 mg Taladegib: 600 mg taladegib administered orally QD on a 28-day cycle.
Arm/Group | 50 mg Taladegib | 100 mg Taladegib | 200 mg Taladegib | 400 mg Taladegib | 600 mg Taladegib
Number analyzed (Participants) | 3 | 6 | 3 | 63 | 7
nanogram*hour/milliliter (μg*h/mL)
  Cycle 1, Day 1 | NA (NA) — For n=3, the minimum=4.07, median=8.87 and maximum=22.1 were reported. | 8.70 (101) | NA (NA) — For n=3, the minimum=8.66, median=12.5 and maximum=50.5 were reported. | 53.7 (99.1) | 96.2 (74.8)
  Cycle 1, Day 15: number analyzed (Participants) | 3 | 6 | 3 | 48 | 2
  Cycle 1, Day 15 | NA (NA) — For n=3, the minimum=7.75, median=7.90 and maximum=72.8 were reported. | 12.4 (113) | NA (NA) — For n=3, the minimum=19.3, median=40.9 and maximum=114 were reported. | 93.8 (103) | NA (NA) — For n=2, individual values 62.6 and 168 were reported.

3. Secondary Outcome: PK: Maximum Observed Drug Concentration (Cmax)
Description: PK: Maximum Observed Drug Concentration (Cmax)
Time Frame: Cycle 1, Day 1: Predose, 0.5, 1, 2, 4, 6, 8, 10,11, 12 hour(h), Day 15: Predose, 0.5, 1, 2, 4, 6, 8, 10,11, 12 h
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | 50 mg Taladegib | 100 mg Taladegib | 200 mg Taladegib | 400 mg Taladegib | 600 mg Taladegib
Number analyzed (Participants) | 3 | 6 | 3 | 63 | 7
microgram per milliliter (μg/mL)
  Cycle 1, Day 1 | NA (NA) — For n=3, the minimum=0.31,median=0.32 and maximum=0.87 were reported. | 0.45 (59.87) | 1.29 (NA) — For n=3, the minimum=1.05,median=1.29 and the maximum=1.43 were reported. | 2.07 (66.39) | 3.28 (34.36)
  Cycle 1, Day 15: number analyzed (Participants) | 3 | 6 | 3 | 48 | 3
  Cycle 1, Day 15 | NA (NA) — For n=3, the minimum=0.30,median=0.38 and maximum=1.36 were reported. | 0.71 (71.67) | NA (NA) — For n=3, the minimum=1.31,median=1.86 and the maximum=2.06 were reported. | 3.62 (59.00) | NA (NA) — For n=3, the minimum=4.85,median=5.94 and maximum=8.23 were collected.

4. Secondary Outcome: PK: Time of Maximal Concentration (Tmax)
Description: PK: Time of Maximal Concentration (Tmax)
Time Frame: Cycle 1, Day 1: Predose, 0.5, 1, 2, 4, 6, 8, 10,11, 12 hour(h), Day 15: Predose, 0.5, 1, 2, 4, 6, 8, 10,11, 12 h
Population: as for outcome 2
Measure: Median (Full Range); unit: hour (h)
Arm/Group | 50 mg Taladegib | 100 mg Taladegib | 200 mg Taladegib | 400 mg Taladegib | 600 mg Taladegib
Number analyzed (Participants) | 3 | 6 | 3 | 63 | 7
hour (h)
  Cycle 1, Day 1 | 2.03 [2.00 to 2.22] | 3.92 [2.00 to 4.00] | 1.22 [0.75 to 4.00] | 2.00 [0.02 to 24.17] | 3.82 [1 to 6]
  Cycle 1,Day 15: number analyzed (Participants) | 3 | 6 | 3 | 48 | 3
  Cycle 1,Day 15 | 2.0 [1.00 to 4.05] | 4.10 [3.78 to 7.80] | 1.00 [0.92 to 1.88] | 2.00 [0.50 to 10.00] | 4.08 [0.88 to 8.00]

5. Secondary Outcome: PK: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC[0-24]) of LSN3185556
Description: PK: Area Under the Plasma Concentration-time Curve from time Zero to 24 Hours (AUC[0-24]) of LSN3185556
Time Frame: Cycle 1, Day 1: Predose, 0.5, 1, 2, 4, 6, 8, 10,11, 12 hour(h), Day 15: Predose, 0.5, 1, 2, 4, 6, 8, 10,11, 12 h
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter (μg*h/mL)
Arm/Group | 50 mg Taladegib | 100 mg Taladegib | 200 mg Taladegib | 400 mg Taladegib | 600 mg Taladegib
Number analyzed (Participants) | 3 | 6 | 3 | 63 | 7
microgram*hour/milliliter (μg*h/mL)
  Cycle 1, Day 1 | NA (NA) — For n=3, minimum=3.46,median=3.85 and maximum=8.95 were reported. | 7.91 (50.1) | NA (NA) — For n=3, the minimum= 14.2, median=17.4 and maximum=28.3 were reported. | 36.6 (70.1) | 67.4 (67.7)
  Cycle 1, Day 15: number analyzed (Participants) | 3 | 6 | 3 | 63 | 2
  Cycle 1, Day 15 | NA (NA) — For n=3, minimum=9.06, median=18.4 and maximum=20.4 were reported. | 22.9 (67.6) | NA (NA) — For n=3, minimum=35.3,median=52.1 and maximum=81.9 were reported. | 121 (81.0) | NA (NA) — n=2, individual values 413 and 465 were reported.

6. Secondary Outcome: PK: Maximum Observed Drug Concentration (Cmax) of LSN3185556
Description: PK: Maximum Observed Drug Concentration (Cmax) of LSN3185556
Time Frame: Cycle 1, Day 1: Predose, 0.5, 1, 2, 4, 6, 8, 10,11, 12 hour(h), Day 15: Predose, 0.5, 1, 2, 4, 6, 8, 10,11, 12 h
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | 50 mg Taladegib | 100 mg Taladegib | 200 mg Taladegib | 400 mg Taladegib | 600 mg Taladegib
Number analyzed (Participants) | 3 | 6 | 3 | 63 | 7
microgram per milliliter (μg/mL)
  Cycle 1, Day 1 | NA (NA) — For n=3, minimum=0.21,median=0.24 and maximum=0.62 were reported. | 0.51 (37.28) | NA (NA) — For n=3, the minimum=0.90,median=1.60 and the maximum=1.71 were reported | 2.27 (62.82) | 4.18 (73.72)
  Cycle 1, Day 15: number analyzed (Participants) | 3 | 6 | 3 | 48 | 3
  Cycle 1, Day 15 | NA (NA) — For n=3, minimum=0.56, median=0.86 and maximum=0.97 were reported. | 1.53 (60.18) | NA (NA) — For n=3, minimum=2.84,median=2.95 and maximum=3.95 were reported | 7.18 (72.20) | NA (NA) — For n=3, minimum= 7.02,median=20.38 and maximum=21.96 were reported.

7. Secondary Outcome: PK: Time of Maximal Concentration (Tmax) of LSN3185556
Description: PK: Time of Maximal Concentration (Tmax)
Time Frame: Cycle 1, Day 1: Predose, 0.5, 1, 2, 4, 6, 8, 10,11, 12 hour(h), Day 15: Predose, 0.5, 1, 2, 4, 6, 8, 10,11, 12 h
Population: as for outcome 2
Measure: Median (Full Range); unit: hour (h)
Arm/Group | 50 mg Taladegib | 100 mg Taladegib | 200 mg Taladegib | 400 mg Taladegib | 600 mg Taladegib
Number analyzed (Participants) | 3 | 6 | 3 | 63 | 7
hour (h)
  Cycle 1, Day 1 | 24.25 [8.00 to 24.48] | 16.81 [6.12 to 24.43] | 6.00 [2.00 to 24.08] | 22.67 [1.13 to 25.17] | 24.00 [7.98 to 24.87]
  Cycle 1,Day 15: number analyzed (Participants) | 3 | 6 | 3 | 48 | 3
  Cycle 1,Day 15 | 8.00 [4.00 to 9.97] | 8.99 [3.78 to 10.00] | 8.00 [8.00 to 24.65] | 1.74 [0.00 to 24.92] | 8.00 [5.82 to 10.17]

8. Secondary Outcome: Number of Participants With Clinical Benefit Rate (Stable Disease [SD] + Partial Response [PR] + Complete Response [CR])
Description: Clinical Benefit Rate is complete response (CR) + partial response (PR) + stable disease (SD) as classified by the investigator according to the Response Evaluation Criteria In Solid Tumors (RECIST version 1.1) guidelines. CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD is a ≥20% increase in the sum of diameter of the target lesions taking as reference the smallest sum on study and an absolute increase in the sum diameter of ≥5 millimeter (mm), the appearance of 1 or more new lesions and/or unequivocal progression of existing nontarget lesions.
Time Frame: Baseline to Disease Progression or Death Due to Any Cause (Up To 32 Months)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Part A: Cohort 3 | Part A: Cohort 4 | Part A: Cohort 5 | Part C | Part D
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 7 | 19 | 40
Participants | 2 | 1 | 2 | 1 | 2 | 4 | 37

9. Secondary Outcome: Part C and D: Progression Free Survival (PFS)
Description: For each participant in Part C and D who is not known to have died or to have had a progression of disease as of the data inclusion cut-off date, PFS was censored at the date of last objective progression-free disease assessment prior to the date of any subsequent systemic anticancer therapy. Progressive disease (PD) was determined using Response Evaluation Criteria In Solid Tumors (RECIST 1.1) criteria. PD is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion.
Time Frame: Baseline to Progressive Disease or Death from Any Cause (Up To 32 Months)
Population: Part C and Part D participants who received at least one dose of study drug and had evaluable PFS data. Participants censored were Part C=8 and Part D=22. Per protocol, Part A data were not collected for PFS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part C | Part D
Number analyzed (Participants) | 11 | 18
months | 1.74 [0.95 to 1.87] | 9.07 [7.36 to NA] — Upper Confidence Interval (CI) was not evaluable due to high censoring.

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly
Arm/Group | Part A: Cohort 1 | Part A: Cohort 2 | Part A: Cohort 3 | Part A: Cohort 4 | Part A: Cohort 5 | Part C | Part D
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/6 | 0/3 | 3/6 | 1/7 | 4/19 | 10/40
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 6/6 | 7/7 | 19/19 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Cohort 1 (N=3) | Part A: Cohort 2 (N=6) | Part A: Cohort 3 (N=3) | Part A: Cohort 4 (N=6) | Part A: Cohort 5 (N=7) | Part C (N=19) | Part D (N=40)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A: Cohort 1 (N=3) | Part A: Cohort 2 (N=6) | Part A: Cohort 3 (N=3) | Part A: Cohort 4 (N=6) | Part A: Cohort 5 (N=7) | Part C (N=19) | Part D (N=40)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (5)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pinguecula (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 5 (5) | 14 (15)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 13 (17)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (3) | 2 (2) | 4 (4) | 8 (9) | 24 (37)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 5 (6) | 3 (5) | 7 (12) | 16 (27)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 3 (3)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 3 (3) | 1 (1) | 2 (2) | 4 (4) | 4 (5) | 9 (9) | 24 (26)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (3)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 21 (23)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 10 (11) | 17 (17)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 3 (4)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Tetany (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Joint lock (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (6) | 2 (2) | 2 (4) | 0 (0) | 1 (1) | 6 (12) | 23 (38)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 11 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 13 (16)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (3) | 3 (3) | 2 (4) | 1 (1) | 4 (4) | 8 (9) | 23 (26)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 7 (13)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Monoplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0/2 (0) | 0/4 (0) | 0/2 (0) | 0/3 (0) | 0/5 (0) | 1/13 (1) | 0/32 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 21 (22)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Part B of the study was not implemented as the estimated half-life was considered long enough for QD dosing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days